CLINICAL TRIAL: NCT02585323
Title: Supporting Physical Activity and Reducing Sedentary Behavior in Arthritis
Brief Title: SuPRA: Using Wearable Activity Trackers With a New Application to Improve Physical Activity in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Simon Fraser University (Other); Arthritis Research Centre of Canada (Other); Fraser Health (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Linda Li, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H15-02038
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Joint Diseases; Knee Osteoarthritis
Keywords: Physical activity; Osteoarthritis; Knee; Exercise; Arthritis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis, Knee; Motor Activity; Osteoarthritis; Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Active Comparator): Education session, Fitbit/FitViz, PT counselling: Participants receive this intervention in Months 1-3. The session will include a presentation on physical activity, an individual goal-setting session with a registered physiotherapist, and an orientation to the Fitbit Flex and the FitViz app. In Months 1 and 2, participants will use the Fitbit/FitViz. The PT will review the progress with participants via 20-minute bi-weekly phone calls, and progressively modify their activities. In Month 3, participants will continue using the Fitbit/FitViz and have access to a PT via email as needed, but no bi-weekly phone calls. In Months 4-9, participants may continue using the Fitbit/FitViz without access to a PT.
  Interventions: Behavioral: Education session, Fitbit/FitViz, PT counselling
- Delayed Intervention Group (Placebo Comparator): Same intervention with a 3 month delay: The full intervention will be initiated in Month 4 and with a brief education session, use of a Fitbit Flex paired with the FitViz app, and counseling by a physiotherapist. In Months 6-9, participants will continue using Fitbit/FitViz without the PT phone calls.
  Interventions: Behavioral: Same intervention with a 3 month delay

INTERVENTIONS:
Behavioral: Education session, Fitbit/FitViz, PT counselling — Participants will receive a brief education session, use a physical activity tracker Fitbit Flex with paired with a FitViz app, and remote counseling by a PT. Intervention will be received immediately.
  Arms: Immediate Intervention Group
Behavioral: Same intervention with a 3 month delay — The Delayed Intervention Group will receive the same intervention as the Immediate Intervention Group, but with a 3 month delay.
  Arms: Delayed Intervention Group

SUMMARY:
Physical activity is an essential first-line treatment for patients with knee osteoarthritis (OA). However, only 13% of patients meet the activity recommendation of 150 minutes or more per week. The primary goal of this randomized controlled trial is to assess the efficacy of a Fitbit Flex (a wireless physical activity tracking device) paired with a new application, plus a brief education session and telephone counselling by a physiotherapist (PT), to improve physical activity and reduce sedentary time in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Current practice guidelines emphasize the use of exercise and weight reduction as the first-line management of knee osteoarthritis (OA; affecting 1 in 10 Canadians). However, up to 90% of people with OA are inactive. Several modifiable risk factors are associated with low physical activity participation, including lack of motivation, doubts about the effectiveness of prescribed exercises and lack of health professional advice regarding ways to progress their physical activity. The variety of risk factors highlights the need for a multifaceted approach that provides support in terms of knowledge, skill development and timely advice from health professionals, as well as motivational support to stay active.

Our primary objective is to assess the efficacy of a Fitbit/Fitviz intervention, involving the use of a Fitbit Flex paired with a FitViz application (app), a brief education session, and telephone counselling by a physiotherapist, to improve physical activity participation and reduce sedentary time in people with knee OA. Our secondary objective is to assess the effect of the intervention on patients' OA disease status and self-efficacy in disease management. We will carry out three aims: 1) To develop the FitViz app to pair with Fitbit to enhance user experience; 2) To conduct a pilot test for the Fitbit/FitViz intervention; 3) To evaluate the effect of the Fitbit/FitViz intervention in patients with knee OA. In this proof-of-concept randomized controlled trial (RCT), the investigators hypothesize that compared to a control group (i.e. the Delayed Intervention Group), participants in the Immediate Intervention Group will 1) increase moderate/vigorous physical activity (MVPA) as determined by an objective measure, 2) reduce sedentary time during waking hours, 3) improve in OA disease status, and 4) improve in their self-efficacy of OA management.

The investigators will use a mixed-method approach, involving a RCT and in-depth interviews. The proof-of-concept study will employ a stepped wedge RCT design, whereby the intervention will be sequentially rolled out to participants over a number of time periods. The order in which individuals receive the intervention will be determined at random. The strength of this design is that it can properly address the efficacy question, while avoiding the dilemma of withholding the intervention to some participants, as in a parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* Have a physician confirmed diagnosis of knee osteoarthritis OR are both 1) over 50, and 2) have experienced 4 weeks of pain, aching, or discomfort in or around the knee during the last year (equal to or more than 28 separate or consecutive days).
* Have no previous diagnosis of inflammatory arthritis (e.g., rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis), connective tissue diseases, or gout.
* Have no history of using disease-modifying anti-rheumatic drugs, such as hydroxychloroquine, sulfasalazine, methotrexate, biologic agents (e.g., Humira, Enbrel), or gout medications.
* Have no prior knee arthroplasty, and not on a waiting list for total knee replacement surgery.
* Have no history of acute injury to the knee in the past 6 months.
* Have not had surgery in the back, hip, knee, or ankle joints in the past 12 months.
* Have an email address and use online/mobile applications.
* Are able to attend one 1.5-hour education session.

Exclusion Criteria:

* Have received a hyaluronate injection in a knee in the last 6 months.
* Have received a steroid injection in a knee in the last 6 months.
* Are at risk when exercising, as identified by the Physical Activity Readiness Questionnaire.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PhD, Principal Investigator — Professor
Locations (1):
- Arthritis Research Canada, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li LC, Feehan LM, Xie H, Lu N, Shaw CD, Gromala D, Zhu S, Avina-Zubieta JA, Hoens AM, Koehn C, Tam J, Therrien S, Townsend AF, Noonan G, Backman CL. Effects of a 12-Week Multifaceted Wearable-Based Program for People With Knee Osteoarthritis: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jul 3;8(7):e19116. doi: 10.2196/19116. PMID 32618578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient participants were recruited between 2017 and 2019 from the Mary Pack Arthritis Program (Vancouver Coastal Health Authority) and the Fraser Health Authority in British Columbia, Canada. We also posted study information on Facebook, Twitter, Kajiji, and Craigslist.
Groups:
- Immediate Intervention Group: Participants received an education session, Fitbit/FitViz, physical therapist (PT) counselling in Weeks 1-13. The session included a presentation on physical activity, an individual goal-setting session with a registered PT, and an orientation to the Fitbit Flex and the FitViz app.
  In Weeks 1-8, participants used the Fitbit/FitViz. The PT reviewed the progress with participants via 20-minute bi-weekly phone calls, and progressively modify their activities.
  In Weeks 9-13, participants continued using the Fitbit/FitViz and had access to a PT via email as needed, but no bi-weekly phone calls.
  In Weeks 14-38, participants did not have access to a PT, but were encouraged to continue using the Fitbit and FitViz.
- Delayed Intervention Group: Participants received the same intervention with a 13-week delay. The full intervention was initiated in Week 14 and with a brief education session, use of a Fitbit Flex paired with the FitViz app, and counseling by a physical therapist (PT).
  In Week 26-38, participants did not have access to a PT but were encouraged to continue using the Fitbit/FitViz.
Period: Baseline
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Started | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 0
Period: Week 13 (RCT Period)
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Started | 26 (Patients) | 25 (Patients)
Completed | 24 (Patients) | 24 (Patients)
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Participant refused assessment | 0 | 1
Period: Week 26 (All Received Intervention)
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Started | 24 (Patients) | 24 (Patients)
Completed | 22 (Patients) | 24 (Patients)
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Week 39 (All Received Intervention)
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Started | 22 (Patients) | 24 (Patients)
Completed | 20 (Patients) | 24 (Patients)
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Immediate Group: Participants received an education session, Fitbit/FitViz, physical therapist (PT) counselling in Weeks 1-13. The session included a presentation on physical activity, an individual goal-setting session with a registered PT, and an orientation to the Fitbit Flex and the FitViz app.
  In Weeks 1-8, participants used the Fitbit/FitViz. The PT reviewed the progress with participants via 20-minute bi-weekly phone calls, and progressively modify their activities.
  In Weeks 9-13, participants continued using the Fitbit/FitViz and had access to a PT via email as needed, but no bi-weekly phone calls.
  In Weeks 14-38, participants did not have access to a PT, but were encouraged to continue using the Fitbit and FitViz.
- Delay Group: Participants received the same intervention with a 13-week delay. The full intervention was initiated in Week 14 and with a brief education session, use of a Fitbit Flex paired with the FitViz app, and counseling by a physical therapist (PT).
  In Week 26-38, participants did not have access to a PT but were encouraged to continue using the Fitbit/FitViz.
- Total: Total of all reporting groups
Arm/Group | Immediate Group | Delay Group | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (8) | 64.8 (9) | 64.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 3 | 6 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 26 | 25 | 51
Daily number of minutes in moderate/vigorous physical activity [Mean (Standard Deviation); unit: Minutes per day] | 31.0 (37.3) | 71.3 (99.8) | 50.8 (76.7)
Daily number of sedentary minutes [Mean (Standard Deviation); unit: Minutes per day] | 567.5 (183.1) | 551.1 (234.9) | 559.4 (208.1)
Daily number of steps [Mean (Standard Deviation); unit: Steps per day] | 6294.0 (3418.0) | 7030.1 (3921.6) | 6654.8 (3655.3)
Knee Injury and Osteoarthritis Outcome Score - Symptom [Mean (Standard Deviation); unit: units on a scale] — The range is 0 to 100, with 0 indicates extreme problems with symptoms and 100 indicates no knee symptoms.
  units on a scale | 68.5 (10.7) | 65.7 (12.3) | 67.2 (11.5)
Knee Injury and Osteoarthritis Outcome Score - Pain [Mean (Standard Deviation); unit: units on a scale] — The range is 0 to 100, with 0 indicates extreme knee pain and 100 indicates no pain.
  units on a scale | 72.6 (13.5) | 65.1 (13.7) | 69.0 (14.0)
Knee Injury and Osteoarthritis Outcome Score - Activity of Daily Living [Mean (Standard Deviation); unit: units on a scale] — The range is 0 to 100, with 0 indicates extreme difficulty with daily tasks and 100 indicates no knee problems and no restriction in daily activities.
  units on a scale | 75.5 (14.7) | 72.2 (15.8) | 73.9 (15.2)
Knee Injury and Osteoarthritis Outcome Score - Sports and Recreation [Mean (Standard Deviation); unit: units on a scale] — The range is 0 to 100, with 0 indicates extreme difficulty and complete inability to participate in sports and recreational activities and 100 indicates perfect knee function with no restrictions.
  units on a scale | 47.9 (23.7) | 46.8 (25.4) | 47.4 (24.3)
Knee Injury and Osteoarthritis Outcome Score - Quality of Life [Mean (Standard Deviation); unit: units on a scale] — The range is 0 to 100, with 0 indicates the worse possible knee problems and 100 indicates no knee problems.
  units on a scale | 44.0 (16.0) | 47.5 (16.0) | 45.7 (17.4)
Partners in Health Scale [Mean (Standard Deviation); unit: units on a scale] — The Partners in Health Scale ranges from 0 to 96, calculated from responses to 12 items on a 9-point Likert scale. A score of 0 represents poor self-management, and a score of 96 represents greater self-management capabilities.
  units on a scale | 76.8 (11.0) | 78.0 (12.0) | 77.4 (11.4)
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 consists of nine questions (rated from 0 to 3) that correspond to nine diagnostic criteria for major depressive disorder. Range 0-27; lower score = less depressive symptoms
  units on a scale | 5.2 (4.6) | 5.4 (5.3) | 5.3 (4.9)
Self-Reported Habit Index - Sitting at Work subscale [Mean (Standard Deviation); unit: units on a scale] | 5.0 (1.4) | 4.5 (2.1) | 4.7 (1.8)
Self-Reported Habit Index - Sitting at Leisure subscale [Mean (Standard Deviation); unit: units on a scale] | 4.8 (1.1) | 5.1 (1.4) | 5.0 (1.2)
Self-Reported Habit Index - Walking subscale [Mean (Standard Deviation); unit: units on a scale] | 4.3 (1.8) | 4.8 (2.0) | 4.5 (1.9)
Theory of Planned Behavior Questionnaire - Attitude toward Physical Activity [Mean (Standard Deviation); unit: units on a scale] | 6.0 (0.6) | 6.1 (0.6) | 6.0 (0.6)
Theory of Planned Behavior Questionnaire - Subjective Norm [Mean (Standard Deviation); unit: units on a scale] | 6.2 (0.6) | 6.3 (0.8) | 6.3 (0.7)
Theory of Planned Behavior Questionnaire - Perceived Control [Mean (Standard Deviation); unit: units on a scale] | 5.8 (1.0) | 6.1 (0.7) | 6.0 (0.9)
Theory of Planned Behavior Questionnaire - Intention [Mean (Standard Deviation); unit: units on a scale] | 6.2 (0.8) | 6.3 (0.8) | 6.3 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Daily Number of Minutes in Moderate/Vigorous Physical Activity
Description: Time spent in Moderate/Vigorous Physical Activity (MVPA) was measured with a SenseWear Mini sensor over a 7-day period. The mean time was calculated in bouted MVPA per day. A bout is defined as >= 10 consecutive minutes or more at the level of >= 3 METs (i.e., the lower bound of MVPA), with allowance for interruption of up to two minutes below the threshold.
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: 13 weeks: Immediate (I) Group: 1 withdrew due to Fitbit wear issues; 1 withdrew, reason unknown. Delayed (D) Group: 1 refused assessment 24 weeks: I Group: 1 withdrew due to family issues, 1 reason unknown 29 weeks: I Group: 2 withdrew - reason unknown
Measure: Mean (Standard Deviation); unit: Minutes per day
Groups:
- Delayed Group: Participants received the same intervention with a 13-week delay. The full intervention was initiated in Week 14 and with a brief education session, use of a Fitbit Flex paired with the FitViz app, and counseling by a physical therapist (PT).
  In Week 26-38, participants did not have access to a PT but were encouraged to continue using the Fitbit/FitViz.
Arm/Group | Immediate Group | Delayed Group
Number analyzed (Participants) | 26 | 25
Minutes per day
  Baseline (T0) | 31.0 (37.3) | 71.3 (99.8)
  13 weeks (T1): number analyzed (Participants) | 24 | 24
  13 weeks (T1) | 37.7 (30.5) | 49.4 (63.6)
  26 weeks (T2): number analyzed (Participants) | 22 | 22
  26 weeks (T2) | 37.0 (32.3) | 74.6 (102.1)
  39 weeks (T3): number analyzed (Participants) | 20 | 23
  39 weeks (T3) | 34.0 (25.2) | 54.8 (66.2)
Statistical Analysis 1: Comparison: Immediate Group vs Delayed Group; We performed an intent-to-treat analysis. For the main comparison, we used analysis of covariance (ANCOVA) to estimate an adjusted mean difference comparing time in MVPA at 13 weeks (primary end point) between groups, adjusting for baseline MVPA, diagnosis, and blocking; Test type: Superiority; p = 0.05, ANCOVA; Adjusted difference in mean change = 13.1, 95% CI 2-sided [1.6 to 24.5]

2. Secondary Outcome: Daily Number of Sedentary Minutes
Description: Time spent in sedentary behaviour was measured with a SenseWear Mini sensor over a 7-day period. The mean daily time spent in sedentary activity was calculated with an energy expenditure of <=1.5 METs, occurring in bouts of >= 20 minutes during waking hours.
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes per day
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
Minutes per day
  Baseline (T0) | 567.5 (183.1) | 551.1 (234.9)
  13 weeks (T1): number analyzed (Participants) | 24 | 24
  13 weeks (T1) | 531.4 (173.5) | 558.3 (224.9)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 492.5 (156.6) | 499.5 (248.9)
  39 weeks (T3): number analyzed (Participants) | 20 | 23
  39 weeks (T3) | 502.8 (135.3) | 483.1 (225.4)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted difference in mean change = -29.5, 95% CI 2-sided [-75.8 to 16.7]

3. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Symptom
Description: The Symptom Subscale ranges from 0 - 100, with 0 indicates extreme knee symptoms and 100 indicates no knee symptoms.
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: 13 weeks: Immediate (I) Group: 1 withdrew due to Fitbit wear issues; 1 withdrew, reason unknown. Delayed (D) Group: 3 refused assessment 26 weeks: I Group: 1 withdrew due to family issues, 1 reason unknown. Delayed (D) Group: 1 refused assessment 39 weeks: I Group: 2 withdrew - reason unknown; 1 refused assessment. Delayed (D) Group: 1 refused assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Group | Delayed Group
Number analyzed (Participants) | 26 | 25
units on a scale
  Baseline (T0) | 68.5 (10.7) | 65.7 (12.3)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 69.3 (12.7) | 66.9 (14.9)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 65.4 (45.8) | 72.2 (16.8)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 68.4 (16.3) | 72.5 (13.3)
Statistical Analysis 1: Comparison: Immediate Group vs Delayed Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted difference in mean change = -1.4, 95% CI 2-sided [-7.8 to 4.9]

4. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Pain
Description: The Pain Subscale ranges from 0 - 100, with 0 indicates extreme knee pain and 100 indicates no knee pain.
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: 13 weeks: Immediate (I) Group: 1 withdrew due to Fitbit wear issues; 1 withdrew, reason unknown. Delayed (D) Group: 3 refused assessment 24 weeks: I Group: 1 withdrew due to family issues, 1 reason unknown. Delayed (D) Group: 1 refused assessment 39 weeks: I Group: 2 withdrew - reason unknown; 1 refused assessment. Delayed (D) Group: 1 refused assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 72.6 (13.5) | 65.1 (13.7)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 73.1 (15.3) | 65.9 (15.6)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 72.5 (18.3) | 74.8 (15.4)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 72.1 (19.8) | 72.8 (13.2)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = 2.5, 95% CI 2-sided [-4.2 to 9.5]

5. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Sport and Recreation
Description: The Sport and Recreation Subscale ranges from 0 - 100, with 0 indicates extreme difficulties with sport and recreational activities due to knee problems and 100 indicates no difficulties.
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
units on a scale
  Baseline (T0) | 47.9 (23.7) | 46.8 (25.4)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 47.1 (22.4) | 52.5 (22.7)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 50.5 (30.1) | 62.5 (22.5)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 51.6 (30.4) | 55.8 (26.3)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = -3.8, 95% CI 2-sided [-14.9 to 7.2]

6. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Activity of Daily Living
Description: The Activity of Daily Living Subscale ranges from 0 - 100, with 0 indicates extreme difficulties with activity of daily living and 100 indicates no difficulties.
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 75.5 (14.7) | 72.2 (15.8)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 75.0 (13.1) | 70.3 (16.9)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 77.7 (18.9) | 80.3 (13.1)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 74.8 (20.7) | 80.0 (14.0)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = 2.8, 95% CI 2-sided [-3.3 to 8.8]

7. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Quality of Life
Description: The Quality of Life Subscale ranges from 0 - 100, with 0 indicates extreme problems with the knee and 100 indicates no problems.
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 44.0 (16.0) | 47.5 (16.0)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 48.7 (17.5) | 46.9 (13.6)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 49.4 (15.7) | 54.7 (14.7)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 49.3 (19.1) | 54.4 (14.6)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = 1.4, 95% CI 2-sided [-5.0 to 7.9]

8. Secondary Outcome: The Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 consists of nine questions (rated from 0 to 3) that correspond to nine diagnostic criteria for major depressive disorder. Range 0-27; lower score = less depressive symptoms),
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 5.2 (4.6) | 5.4 (5.3)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 4.0 (3.0) | 4.7 (4.9)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 3.6 (3.3) | 4.5 (5.2)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 4.2 (4.1) | 4.5 (5.3)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = -0.4, 95% CI 2-sided [-1.7 to 0.8]

9. Secondary Outcome: Partners in Health Scale
Description: The Partners in Health Scale ranges from 0 to 96, calculated from responses to 12 items on a 9-point Likert scale. A score of 0 represents poor self-management, and a score of 96 represents greater self-management capabilities.
Time Frame: Baseline, Months 3, 6, and 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 76.8 (11.0) | 78.0 (12.0)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 76.7 (11.5) | 81.6 (9.6)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 78.9 (9.0) | 82.6 (9.3)
  29 weeks (T3): number analyzed (Participants) | 19 | 24
  29 weeks (T3) | 81.0 (7.0) | 82.6 (10.0)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = -2.3, 95% CI 2-sided [-6.6 to 1.9]

10. Secondary Outcome: Self-Reported Habit Index (SRHI) - Sitting at Work Subscale
Description: The SRHI is a 12-item scale, rated on a 7-point Likert scale, that measures characteristics of habitual behavior. In the Habit index, participants rated their strength of habit for three specific activity-related behaviors: sitting during leisure time at home, sitting during usual occupational activities, and walking outside for 10 minutes. A higher score indicates a stronger habit or behavior that is done frequently, automatically, and done without thinking about it. Range 1-7; higher score = stronger habit.
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 5.0 (1.4) | 4.5 (2.1)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 5.2 (1.6) | 4.4 (2.0)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 4.7 (2.1) | 4.3 (2.1)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 5.0 (1.9) | 4.1 (2.1)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = 0.7, 95% CI 2-sided [0.2 to 1.2]

11. Secondary Outcome: Self-Reported Habit Index (SRHI) - Sitting at Leisure Subscale
Description: as for outcome 10
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 4.8 (1.1) | 5.1 (1.4)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 5.1 (1.1) | 4.7 (1.6)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 5.0 (1.1) | 4.4 (1.9)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 5.5 (1.1) | 4.7 (1.7)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = 0.7, 95% CI 2-sided [0.2 to 1.1]

12. Secondary Outcome: Self-Reported Habit Index (SRHI) - Walking Subscale
Description: as for outcome 10
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 4.3 (1.8) | 4.8 (2.0)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 4.4 (1.6) | 4.6 (2.0)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 4.6 (1.8) | 4.8 (1.6)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 4.7 (1.8) | 4.6 (1.8)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = 0.3, 95% CI 2-sided [-0.3 to 0.9]

13. Secondary Outcome: Theory of Planned Behavior Questionnaire - Attitude Toward Physical Activity
Description: The Theory of Planned Behavior Questionnaire consists of 16 items measuring all components of theory. It was used to measure motivation for physical activity. Range: 1-7; higher = more positive)
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 6.0 (0.6) | 6.1 (0.6)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 5.9 (0.7) | 6.1 (0.7)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 6.0 (0.5) | 6.2 (0.6)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 6.0 (0.5) | 6.1 (0.7)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = -0.1, 95% CI 2-sided [-0.4 to 0.2]

14. Secondary Outcome: Theory of Planned Behavior Questionnaire - Subjective Norm
Description: as for outcome 13
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 6.2 (0.6) | 6.3 (0.8)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 6.2 (0.8) | 6.2 (0.7)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 6.1 (0.8) | 6.3 (0.8)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 6.2 (1.1) | 6.3 (0.7)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = 0.2, 95% CI 2-sided [-0.1 to 0.5]

15. Secondary Outcome: Theory of Planned Behavior Questionnaire - Perceived Control
Description: as for outcome 13
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 5.8 (1.0) | 6.1 (0.7)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 5.6 (1.4) | 5.8 (1.2)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 5.6 (1.5) | 6.2 (1.0)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 5.7 (1.4) | 6.2 (0.9)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = 0.1, 95% CI 2-sided [-0.6 to 0.8]

16. Secondary Outcome: Theory of Planned Behavior Questionnaire - Intention
Description: as for outcome 13
Time Frame: Baseline, 13 weeks, 26 weeks, 39 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 26 | 25
score on a scale
  Baseline (T0) | 6.2 (0.8) | 6.3 (0.8)
  13 weeks (T1): number analyzed (Participants) | 24 | 22
  13 weeks (T1) | 5.9 (1.0) | 6.4 (0.6)
  26 weeks (T2): number analyzed (Participants) | 22 | 24
  26 weeks (T2) | 5.7 (1.1) | 6.3 (0.6)
  39 weeks (T3): number analyzed (Participants) | 19 | 24
  39 weeks (T3) | 5.8 (0.8) | 6.3 (0.9)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; Test type: Superiority; p = 0.05, ANCOVA; Adjusted diff in mean change at T0-T1 = 0.1, 95% CI 2-sided [-0.1 to 0.3]

ADVERSE EVENTS:
Time Frame: 39 weeks
Description: Self-reported adverse events were collected, including cardiovascular events, musculoskeletal events (e.g., muscle pain, ligament sprain), or falls while being physically active, were collected.
Groups:
- Immediate Group: Education session, Fitbit/FitViz, PT counselling: Participants received this intervention in Weeks 1-13. The session included a presentation on physical activity, an individual goal-setting session with a registered physiotherapist, and an orientation to the Fitbit Flex and the FitViz app. In Weeks 1-8, participants used the Fitbit/FitViz. The PT reviewed the progress with participants via 20-minute bi-weekly phone calls, and progressively modify their activities. In Weeks 9-13, participants continued using the Fitbit/FitViz and had access to a PT via email as needed, but no bi-weekly phone calls.
  In Weeks 14-38, participants did not have access to a PT, but were encouraged to continue using the Fitbit/FitViz.
- Delay Group: Same intervention with a 13-week delay: The full intervention was initiated in Week 14 and with a brief education session, use of a Fitbit Flex paired with the FitViz app, and counseling by a physiotherapist.
  In Week 26-38, participants did not have access to a PT, but were encouraged to continue using the Fitbit/FitViz.
Arm/Group | Immediate Group | Delay Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 7/26 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Group (N=26) | Delay Group (N=25)
Fall during physical activity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
With the use of a delay-control design in which the participants in the control arm received the program after a 13-week delay, the efficacy of the program could only be unequivocally assessed at 13 weeks. The results may not be generalizable to men because 82% of the participants were women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT02585323/Prot_SAP_000.pdf